CLINICAL TRIAL: NCT03572959
Title: Management of Pain in Oral Lichen Planus Patients: A Comparative Pilot Study
Brief Title: Management of Pain in Oral Lichen Planus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sherine Adel Nasry (Other)
Responsible Party: Sponsor-Investigator, Sherine Adel Nasry, Associate Professor, National Research Centre, Egypt
Organization: National Research Centre, Egypt (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 15023
Record Dates: First submitted 2018-06-19; First posted 2018-06-28 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Oral Lichen Planus
MeSH Terms: conditions — Lichen Planus, Oral | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- comparison group (active control) (Active Comparator): 0.1 % topical triamcinolone acetonide preparation (Kenacourt-A Orabase Pomad, DEVA HOLDINGS A.S., Istanbul, Turkey) was used where the patients' were instructed to apply the gel 4 times daily, with no food or fluid taken one hour after application. Patients used the medication for 4 weeks , and if extension of treatment was required after that period , patients were instructed to apply miconazole oral gel (JANSSEN-CILAG Pty Ltd 1-5 Khartoum Road North Ryde NSW 2113 Australia) four times a day for one week to protect from superimposed fungal infections.15
  Interventions: Drug: 0.1 % topical triamcinolone acetonide
- experimental group (Experimental): OLP lesions were irradiated with a 970-nm diode laser (SIRO Laser Advance class III b, SIRONA, Germany) with a 2 W irradiation power in a continuous non-contact mode. The laser beam was delivered using a fiber-optic tip with a 320 µm diameter with defocused mode directed at the lesions plus 0.5 cm peri- lesional tissues with a slight overlapping in order to evenly distribute energy covering all the lesional and peri-lesional tissues until blanching of the area was observed.14 Diode laser was calibrated to an output power of 3W, frequency of 30 Hz, energy of 180 joule and time interval of 8 minutes divided into 4 sessions , two min each with one minute rest in between to allow for tissue relaxation.
  Irradiation was done twice weekly for two months until the resolution of signs for a maximum of ten sessions.11 After each session, patients were advised to have a cold diet and use chlorhexidine oral gel postoperatively twice a day to the lesion for one week.
  Interventions: Device: SIROIaser

INTERVENTIONS:
Drug: 0.1 % topical triamcinolone acetonide — 0.1 % topical triamcinolone acetonide preparation was used where the patients' were instructed to apply the gel 4 times daily, with no food or fluid taken one hour after application.
  Arms: comparison group (active control)
Device: SIROIaser — Oral Lichen Planus lesions were irradiated with a 970-nm diode laser with a 2 W irradiation power in a continuous non-contact mode. The laser beam was delivered using a fiber-optic tip with a 320 µm diameter with defocused mode directed at the lesions plus 0.5 cm peri- lesional tissues with a slight overlapping in order to evenly distribute energy covering all the lesional and peri-lesional tissues until blanching of the area was observed.14 Diode laser was calibrated to an output power of 3W, frequency of 30 Hz, energy of 180 joule and time interval of 8 minutes divided into 4 sessions , two min each with one minute rest in between to allow for tissue relaxation.
  Irradiation was done twice weekly (once every third day) for two months until the resolution of signs for a maximum of ten sessions.
  Arms: experimental group

SUMMARY:
Treating Oral Lichen Planus (OLP) is a big challenge for clinicians. Despite numerous existing remedies, to date no effective cure has been found, which is mainly attributed to the lack of understanding of the pathogenesis of the disease. The investigator's aim was comparing the effectiveness of topical steroids and diode laser in treating OLP patients. Twenty-four patients with OLP were allocated into two groups of twelve patients each. One group was treated with 970 nm diode laser applied twice weekly and the other group was treated with topical steroids applied four times per day. Patients were followed up for two months. Pain was recorded using the visual analog score (VAS) and the clinical signs and symptoms were recorded using the reticular, atrophic, erosive (RAE) sores. Pain and RAE records were taken before treatment, after treatment and after 2 months.

DETAILED DESCRIPTION:
24 patients (16 females , 8 males ) were recruited in this study from the Dental Clinic of the National Research Centre, Egypt, and the Ethical Committee approved the study protocol. All patients were informed about the treatment plan and they all submitted a written informed consent before enrolment, which was carried out in accordance with the declaration of Helsinki. Inclusion criteria included oral lesions clinically and histopathologically consistent with the modifications for the WHO 2003 criteria suggested by van der Meij and van der Waal.13 Patients were excluded from the study in case of indefinite diagnosis (such as lichenoid inflammation); or those suffering from any disease that may present with features similar to OLP (graft versus host disease or lupus erythematosus),if they received any medication for OLP treatment in the two months prior enrolment in the study, if they were pregnant or lactating women, or if histological diagnosis revealed lichenoid changes or any signs of dysplasia. 4,14

Study design:

Patients were randomly divided into two groups using a randomization software, where a blocked randomization was used to ascertain equal distribution of patients into each group (parallel-group study).15 One group (12 patients) was irradiated with diode laser and the other group was treated with topical steroids. In the laser group, normal protective measures were taken, where patients and personnel wore laser safety glasses . OLP lesions were irradiated with a 970-nm diode laser (SIRO Laser Advance class III b, SIRONA, Germany) with a 2 W irradiation power in a continuous non-contact mode. The laser beam was delivered using a fiber-optic tip with a 320 µm diameter with defocused mode directed at the lesions plus 0.5 cm peri- lesional tissues with a slight overlapping in order to evenly distribute energy covering all the lesional and peri-lesional tissues until blanching of the area was observed.14 Diode laser was calibrated to an output power of 3W, frequency of 30 Hz, energy of 180 joule and time interval of 8 minutes divided into 4 sessions , two min each with one minute rest in between to allow for tissue relaxation.

Irradiation was done twice weekly (once every third day) for two months until the resolution of signs (meaning the resolution of all atrophic-erosive lesions, regardless of any persisting hyperkeratotic lesions) for a maximum of ten sessions.11 After each session, patients were advised to have a cold diet and use chlorhexidine oral gel postoperatively. The patients applied the gel twice a day to the lesion for one week.16 For the steroid group (12 patients), 0.1 % topical triamcinolone acetonide preparation (Kenacourt-A Orabase Pomad, DEVA HOLDINGS A.S., Istanbul, Turkey) was used where the patients' were instructed to apply the gel 4 times daily, with no food or fluid taken one hour after application. Patients used the medication for 4 weeks , and if extension of treatment was required after that period , patients were instructed to apply miconazole oral gel (JANSSEN-CILAG Pty Ltd 1-5 Khartoum Road North Ryde NSW 2113 Australia) four times a day for one week to protect from superimposed fungal infections.15 Scoring of the clinical signs was done according to the RAE (Reticular, Erosive, Atrophic ) scale of Thongprasom and co- workers.17 Total improvement of the clinical signs was given scores zero or one and was defined as the disappearance of all atrophic-erosive lesions, whether any hyperkeratotic lesions persisted or not. Partial improvement or persisting of the patient's condition meant a decrease (score 2, 3 or 4), or no improvement (no change in the patient's score). Hence the clinical and symptomatic improvement of the patient's lesion was expressed by the numerical difference between baseline and endpoint scores. 14 Pain was recorded using the Visual Analogue Scale (VAS), which consisted of a 10-cm horizontal line, starting from 0 (designating no pain experienced by the patient to 10 (designating unbearable or most severe pain). Pain and RAE records were taken before treatment, after treatment and then after 2 months follow up.

ELIGIBILITY:
Inclusion Criteria:

* histological diagnosis of OLP on the basis of WHO criteria (Meji and van der Waal 2003).
* presence of painful and atrophic-erosive oral lesions, unresponsive to topical corticosteroid therapy
* ability to complete the present clinical trial.

Exclusion Criteria:

* Presence of histological signs of dysplasia
* use of lichenoid reaction inducing drugs
* Therapy for OLP in the 2 months prior to the study;
* Patients suffering from any disease that may present with features similar to OLP (graft versus host disease or lupus erythematosus)
* Pregnant or lactating females
* Patients with uncontrolled diabetes or hypertension, positive HCV Ab or HBs Ag.
* Smokers

Ages: 45 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-12-27 (Actual); Primary Completion 2017-03-20 (Actual); Study Completion 2017-05-22 (Actual)

PRIMARY OUTCOMES:
change in VAS | two months
  Visual Analogue Scale (VAS) The pain VAS is a continuous single-item scale comprised of a horizontal (HVAS) or vertical (VVAS) line, usually 10 centimeters in length, anchored by 2 verbal descriptors, one for each symptom extreme Range: 0-10 (cm) no pain (0-0.4 cm), mild pain (0.55-4.4 cm), moderate pain (4.5-7.4)cm, and severe pain (7.5- 10) cm A higher score indicates greater pain intensity

SECONDARY OUTCOMES:
change in RAE | two months
  The Reticular, Atrohpic, Erosive ( RAE ) scale used by Thongprasom and co-workers records and measures the clinical appearance of the Oral Lichen Planus) OLP lesion Score range: 0-5 with o being the most favorable clinical appearance and 5 the most severe clinical appearance.
  score 0: no lesions; score 1: hyperkeratotic lesions score 2: atrophic area ≤1 cm2 score 3: atrophic area >1 cm2 score 4: erosive area ≤1 cm2 score 5: erosive area >1 cm2

IPD SHARING:
Plan to Share IPD: No